CLINICAL TRIAL: NCT00844675
Title: Effects of Preoperative Administration of Oral Rabeprazole on the Prevention of Ulcer Bleeding Following Endoscopic Mucosal Resection(EMR): Prospective, Randomized, Placebo-controlled, Comparative Study
Brief Title: Effects of Oral Rabeprazole on the Prevention of Ulcer Bleeding Following Endoscopic Mucosal Resection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Catholic University of Korea (Other)
Collaborators: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Principal Investigator, Myung-gui Choi, MD, PhD, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RAB-KOR-9035
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2012-10-18 (Estimated); Status verified 2012-10

CONDITIONS: Early Gastric Adenocarcinoma; Adenocarcinoma, Tubular
Keywords: endoscopic mucosal resection; Proton Pump Inhibitor; gastrointestinal hemorrhage; rabeprazole
MeSH Terms: conditions — Adenocarcinoma; Gastrointestinal Hemorrhage | interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rabeprazole (Experimental): rabeprazole
  Interventions: Drug: rabeprazole
- placebo (Experimental): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rabeprazole — The rabeprazole group will receive oral rabeprazole 20mg twice day (morning and evening) 30 minutes before meals from 5 days before EMR (D-5) to 1 day before EMR (D-1).
  Other Names: Pariet(rabeprazole)
  Arms: rabeprazole
Drug: placebo — The placebo group will receive a placebo by mouth twice a day (morning and evening) 30 minutes before meals from 5 days before EMR (D-5) to 1 day before EMR (D-1).
  Arms: placebo

SUMMARY:
The purpose of this study is:

* To examine if oral administration of Pariet (proton pump inhibitor, 20mg tablets, twice daily for 5 days) before Endoscopic mucosal resection(EMR) exhibits preventive effects of ulcer bleeding compared with placebo group (preoperative administration of placebo)
* To evaluate the effects on the suppression of acid secretion of preoperative administration of an Proton pump inhibitor

DETAILED DESCRIPTION:
* Endoscopic mucosal resection (EMR) is less invasive than surgery and is known to be general treatment for early gastric cancer or gastric adenoma when patients' quality of life is taken into consideration. However, major complications such as bleeding and perforation remain to be problematic.1-5 The incidence of these complications is expected to rise as the size of lesions for which EMR is indicated has enlarged. Histamine 2 receptor antagonists (H2RA) and proton pump inhibitors (PPI) have been used for the bleeding,1-3 but the bleeding rate following EMR has been reported to be still high as 1.4% to 24%.1,4 Green et al and Berstad et al cited in their research that intragastric PH should be sustained above 5.4 to prevent bleeding, and PPIs should be administered instead of H2RAs to keep PH above 5.4. Being studied are administration modalities to enhance the therapeutic efficacy of PPIs or H2RAs.1-3 Several studies have already demonstrated that high-dose PPI therapy, for which a PPI was administered twice daily, effectively blocks acid secretion by increasing intragastric pH to neutral.3 Our study team also suggested in a previous study that high-dose PPI therapy was adequate to maintain intragastric pH above 6.
* PPIs are known to induce the suppression of acid secretion because they destroy a proton pump, yet it takes 5 days to achieve their maximum effects.7,8 It's been suggested that the onset of PPIs is slow to prevent bleeding with administration of a PPI after EMR.4 Therefore, our investigators expect that 5-day administration of an oral PPI before EMR would increase intragastric pH to above 6 and would be at least equal to or superior to intravenous PPIs currently being used in terms of the suppression of acid secretion.
* This is a prospective, randomized, comparative study to substantiate that oral administration of rabeprazole (Pariet tablets) 20mg twice daily before and after EMR (PO RBP group) will show similar effects on the prevention of bleeding compared with the conventional treatment with iv administration of pantoprazole after EMR but no special medication given before EMR (Placebo group). In addition, we are going to measure intragastric pH among part of study subjects and then to evaluate if the effect of acid suppression in the PO RBP group is superior to that in the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have EMR planned as well as meet the criteria described below will be selected as study subjects
* Patients in whom EMR is indicated:

  1. Gastric adenoma
  2. Early gastric adenocarcinoma

     * Moderately or well differentiated adenocarcinoma
     * Gastric cancer limited to only mucosa on endoscopic ultrasonography
     * No invasion of lymph nodes or metastases (diagnosed by CT)
  3. EMR to be performed for other diagnostic purposes
* Women of child-bearing potential should avoid pregnancy
* Subjects who consented to a EMR procedure in writing

Exclusion Criteria:

* Patients who meet the criteria described below should be excluded from study subjects:

  1. Younger than 18 years old
  2. Patients with a history of upper gastrointestinal surgery or vagotomy
  3. Patients with serious adverse reactions secondary to cardiac, renal, hepatic, or hematologic diseases (e.g. creatinine> 2.5 mg/dl, total bilirubin >3.0 mg/dl)
  4. Patients with diseases that may have a great impact on the clinical study
  5. Patients to whom the stimulation of gastrointestinal movement poses risks as in gastrointestinal bleeding, mechanical ileus and perforation
  6. Women who are pregnant or nursing
  7. Patients who are being treated with adrenocorticoid steroids, nonsteroidal anti-inflammatory drugs including aspirin, or other ulcer inducers
  8. Patients who are taking other antiulcer drugs (antacids, antihistamines, etc) that may affect the efficacy assessments of the study drug (but, except for patients not taking the drugs over 7 days)
  9. Patients with severe psychiatric diseases
  10. Patients who received other investigational drugs within 30 days prior to the start of this study or who are currently participating in other clinical study
  11. Patients who did not consent to the clinical study
  12. Patients who can not be examined
* Patients with bleeding tendency
* Patients with esophageal varices
* Patients with esophageal ulcer, stricture, or obstruction
* Patients who have pacemaker or implantable cardiac defibrillator in place

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-10; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Frequency of bleeding after EMR is performed | 4weeks

SECONDARY OUTCOMES:
Number (No./cm2) of visible vessels on the fundus of ulcer on endoscopy performed within 24 hours after EMR | day 1
Percentage of a pH change with intragastric pH greater than 6 in 24 hours after EMR | day 0
Measurement of a change in the size of ulcer | 4weeks

CONTACTS AND LOCATIONS:
Overall Officials: MyungKu Choi, MD, Principal Investigator — The Catholic University of Korea
Locations (1):
- Catholic University, Gangnam St. Mary's Hospital, Seoul, Ban-po Dong 505, South Korea